CLINICAL TRIAL: NCT01492673
Title: A Phase II Trial of Cyclophosphamide, Topotecan, and Bevacizumab (CTB) in Patients With Relapsed/Refractory Ewing's Sarcoma and Neuroblastoma
Brief Title: Cyclophosphamide, Topotecan, and Bevacizumab (CTB) in Patients With Relapsed/Refractory Ewing's Sarcoma and Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Children's Mercy Hospital Kansas City (Other); Penn State University (Other); University of Colorado, Denver (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other); Phoenix Children's Hospital Center for Cancer & Blood Disorders (Unknown); Alberta Children's Hospital (Other); MD Anderson Cancer Center Orlando (Unknown); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-183
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2018-10

CONDITIONS: Neuroblastoma; Sarcoma
Keywords: Ewing's sarcoma; BEVACIZUMAB (AVASTIN); CYCLOPHOSPHAMIDE (CYTOXAN); TOPOTECAN; 11-183; POETIC
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Sarcoma, Ewing | interventions — Cyclophosphamide; Topotecan; Bevacizumab

ARMS (1):
- Cyclophosphamide, Topotecan, and Bevacizumab (CTB) (Experimental): This is a multi-center, open label phase II study evaluating the safety and efficacy of the novel combination of agents consisting of bevacizumab, cyclophosphamide, and topotecan.
  Interventions: Drug: Cyclophosphamide, Topotecan, and Bevacizumab

INTERVENTIONS:
Drug: Cyclophosphamide, Topotecan, and Bevacizumab — The treatment schedule for this study will consist of a 21-day cycle. Dose modification will only occur with administration of the investigational agent, bevacizumab. The schedule of administration is summarized as follows. Administration of bevacizumab will precede the administration of the cyclophosphamide and topotecan by 3 days (Day - 3) to allow for vascular stabilization prior to initiation of chemotherapy. The chemotherapy backbone will consist of cyclophosphamide and topotecan administered as follows: cyclophosphamide 250 mg/m2/day IV over 30 minutes ± 5 minutes on Days 0-4 followed by topotecan 0.75 mg/m2/day IV over 30 minutes ± 5 minutes on Day 0-4 of every cycle. The dosing of cyclophosphamide and topotecan will be fixed.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad treatment with a new combination of drugs, cyclophosphamide, topotecan, and bevacizumab has on the patient and their cancer.

The medications, cyclophosphamide and topotecan, are standard drugs often used together for the treatment of cancer in children with either Ewing's sarcoma or neuroblastoma.

Bevacizumab is an experimental drug called an antibody that targets a protein important in the growth of cancer cells called vascular endothelial growth factor (VEGF). VEGF is made by tumor and other surrounding cells to help make blood vessels needed for the growth and spread of cancer cells in the body. The way that bevacizumab works is to stop the cancer cells from making their own blood supply, causing the tumor to stop growing bigger or from spreading. In adult clinical trials, bevacizumab has shown promising anti-cancer activity in patients with cancer of the colon/rectum (colorectal) and breast. It has been approved by the Food and Drug Administration (FDA) for use in patients with colorectal cancer but not in cancers found in children. Bevacizumab has been tested in early clinical studies in children and has been shown to be safe.

Other goals of this study will include research tests designed to test the following changes in the patient or their cancer: to see how the body handles and breaks down bevacizumab (pharmacokinetics), to look at changes in proteins in the blood that may affect the way the cancer responds to the combination (angiogenic profile, angiogenesis associated serum biomarkers), to look at changes in genes that may affect how the cancer responds to treatment with this combination of medications (metabolic signature), and to monitor the effects of changes in the way the body grows and develops before and after bevacizumab is given.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed/refractory Ewing's sarcoma or neuroblastoma.
* Patients must have measurable disease. Patients with a diagnosis of neuroblastoma with MIBG avid disease only are permitted to enroll on this study.
* Patients must be ≤ 21 years of age at time of diagnosis
* Life expectancy ≥ 3 months
* Lansky or Karnofsky performance ≥ 70%
* Written informed consent
* Organ and marrow function defined as follows:

Hematologic function, as follows

* Absolute neutrophil count ≥ 1000/μL
* Platelets ≥ 100 x 109/L (without transfusion < 14 days before enrollment) Hemoglobin ≥ 9 gm/dl

Renal function, as follows:

* Serum creatinine ≤ ULN for age. Refer to Appendix H for normal values for serum creatinine in children.
* If serum creatinine above these values, the calculated creatinine clearance or radioisotope GFR must be ≥ 60 ml/min/1.73 m2
* Urinary protein < 2+ (unless total quantitative protein is < 500 mg protein/day as determined by 24 H urine collection) for pediatric patients please refer to the CTCAE V4.0 for values.

Hepatic function, as follows:

* Total bilirubin ≤ 1.5x ULN
* AST and ALT ≤ 2.5x ULN for institution or ≤ 5x ULN for institution if clearly attributable to liver metastases
* Albumin ≥ 2.5 g/dl. Coagulation: INR ≤ 1.5x ULN.
* Prior Treatment: Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiation therapy prior to entry on study. Patients must have had at least one prior treatment regimen. Patients may have received treatment previously with cyclophosphamide or topotecan but no prior bevacizumab.
* Myelosuppressive chemotherapy: Two weeks must have elapsed since administration of previous chemotherapy.
* Biologic agents: At least 2 weeks must have elapsed since the completion of therapy with a monoclonal antibody. Seven days must have elapsed since the last dose of retinoids
* Radiation therapy: For all patients, ≥ 4 weeks must have elapsed for local XRT; ≥ 6 months must have elapsed if prior radiation to ≥ 50% of the pelvis or if substantial bone marrow irradiation. Patients with a history of prior radiation with field including the heart (e.g. mantle) will be excluded.
* Stem cell transplant: Patients who have undergone prior stem cell transplantation will not be excluded from study entry. At least 3 months must have elapsed since autologous or allogeneic stem cell transplantation. Patients must have no evidence of active graft versus host disease.

Exclusion Criteria:

* Patients with centrally-located pulmonary or mediastinal primary tumors or metastases adjacent to or invading large blood vessels.
* Prior left chest wall irradiation or a cumulative anthracycline dose of greater or equal to 300 mg/m2, unless the ejection fraction or fraction shortening is within normal institutional limits, in which case the patient can be enrolled.
* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 3 months
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Active second malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years
* History of other malignancies, except for other solid tumors curatively treated with no evidence of disease for > 3 years prior to enrollment.
* Known infection with human immunodeficiency virus (HIV).
* Uncontrolled hypertension (sBP >150 mmHg and/or diastolic BP > 100 mmHg, found on two consecutive measurements separated by a one week period of time despite adequate medical support).
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day - 3.
* History of stroke or transient ischemic attack within 6 months prior to Day -3.
* Known CNS disease, except for treated brain metastases.
* Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day -3 will be excluded.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day -3.
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day -3.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day -3 or anticipation of need for major surgical procedure during the course of the study. (A major procedure constitutes an invasive procedure which requires general anesthetic support, hospitalization, and supportive care such as laparotomy, laminectomy, etc.)
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1. (Minor surgical procedures include minimally invasive procedures such as fine needle aspiration, core biopsy, etc requiring little if any supportive care excluding lumbar puncture and bone marrow aspiration/biopsy.)
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day -3.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Thrombolytics or treatment doses of warfarin within 28 days of initiating treatment. Patients who require low dose warfarin for central venous catheter patency are allowed to enter if their dose is < 2 mg per day total AND their International Normalized Ratio (INR) is ≤ 1.5.
* Patients requiring treatment doses of heparin for any reason. The use of heparin flushes for maintenance of central venous catheters is permitted
* Patients requiring aspirin > 325 mg per day or non-steroidal anti-inflammatory medications known to inhibit platelet function. Patients taking cyclooxygenase-2 inhibitors (COX-2) inhibitors are allowed to enroll.
* History or clinical evidence of deep venous thrombosis including pulmonary embolus within 6 months of treatment.
* Patients with proteinuria > 1+ on urine dipstick or UPC ratio ≥ 1.0 at screening. If >1+ proteinuria is detected on surveillance, a 24-hour collection must be performed if eligibility is desired. Patients with a 24-hour urine protein content of ≤ 500 mg are eligible.
* Known hypersensitivity to any component of bevacizumab.
* Pregnancy (positive pregnancy test) or lactation. (An effective means of contraception (men and women) in subjects of child-bearing potential must be used.)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (6):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - University of Colorado Health Sciences Center and The Children's Hospital, Denver, Colorado
  - MD Anderson Cancer Center Orlando at Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
- Alberta Children'S Hospital, Calgary, Alberta, Canada

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclophosphamide, Topotecan, and Bevacizumab (CTB)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, Topotecan, and Bevacizumab (CTB)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 12 [8 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: as measured by objective response rate (CR/PR) after 2 cycles of treatment and duration of response. after 2 cycles of treatment and duration of response according to the Revised RECIST guideline (version 1.1)
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: Data were not collected. Study terminated due to low accrual.
Arm/Group | Cyclophosphamide, Topotecan, and Bevacizumab (CTB)
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety will be assessed by physical examination, interim history, and laboratory assessments. Adverse events will be graded according to the NCI-CTCAE, version 4.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, Topotecan, and Bevacizumab (CTB)
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cyclophosphamide, Topotecan, and Bevacizumab (CTB)
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Topotecan, and Bevacizumab (CTB) (N=9)
Alanine aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 1
Oral pain (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 7
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
White blood cell decreased (Investigations) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Topotecan, and Bevacizumab (CTB) (N=9)
Anemia (Blood and lymphatic system disorders) | 7
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 7
White blood cell decreased (Investigations) | 7
Nausea (Gastrointestinal disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Headache (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT01492673/Prot_SAP_000.pdf